CLINICAL TRIAL: NCT06433180
Title: A Prospective, Multi-center, Double Blind Randomized Trial of Fecal Microbiota Transplantation (FMT) Delivered by Capsule Versus Placebo in Severe Irritable Bowel Syndrome (IBS).
Brief Title: Study of Fecal Microbiota Transplantation (FMT) in Severe IBS Patients
Acronym: ICEBOAT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP180583; 2019-003433-41 (EudraCT Number)
Record Dates: First submitted 2024-05-13; First posted 2024-05-29 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: fecal microbiota transplantation; irritable bowel syndrome; frozen capsule; Rome IV; IBS-SSS
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Administration of the sham (PLACEBO) (Placebo Comparator): Oral, capsulized, frozen capsules without fecal matter but containing cryopreservation solution will be administered at the same volume and same time point as in the experimental group. Taken in one day in two separate meals. Administration of the sham after colon cleaning.
  Interventions: Drug: Administration of the sham (PLACEBO)
- Administration of fecal microbiota transplantation ( FMT capsules) (Experimental): Oral, capsulized, frozen fecal microbiota transplantation FMT delivering approximatively 24 g of stools taken in one day in two separate meals. Administration of the FMT after colon cleaning.
  Interventions: Drug: Administration of fecal microbiota transplantation ( FMT capsules)

INTERVENTIONS:
Drug: Administration of fecal microbiota transplantation ( FMT capsules) — Oral, capsulized, frozen fecal microbiota transplantation FMT delivering approximatively 24 g of stools taken in one day in two separate meals. Administration of the FMT after colon cleaning.
  Arms: Administration of fecal microbiota transplantation ( FMT capsules)
Drug: Administration of the sham (PLACEBO) — Oral, capsulized, frozen capsules without fecal matter but containing cryopreservation solution will be administered at the same volume and same time point as in the experimental group. Taken in one day in two separate meals. Administration of the sham after colon cleaning.
  Arms: Administration of the sham (PLACEBO)

SUMMARY:
The objective of this protocol is to evaluate the efficacy of fecal microbiota transplantation (FMT) using oral capsules containing frozen stools vs sham FMT on IBS severity score at 12 weeks in patients with severe irritable bowel syndrome refractory to conventional treatments.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a chronic disease. It affects about 4.4 to 10 % of the French general population (according to Rome III or Rome IV definition) and is the most frequent functional bowel disorder in patients visiting general practitioners or gastroenterologists. The efficacy of treatments is often limited, in particular form the case severe of IBS (IBS-SSS>300) which concerns at least 20 to 25% of patients and IBS can cause significant deterioration in quality of life.

In this context, microbiota could become a potential therapeutic target, and replacement of the abnormal fecal microbiota by an "healthy" one, especially in patients refractory to previous treatment and with severe symptoms, is a seducing new therapeutic strategy. The primary outcome is an improvement in the IBS-SSS score level at 12 weeks after taking a oral capsules of FMT in patients with severe IBS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and < 75 years
* IBS defined according to Rome IV definition (IBS-C, IBS-D or IBS-M)
* Severe disease (IBS-SSS >300) and refractory to at least two previous treatment strategies:among the following : anti-spasmodic and/or laxatives (polyethylene glycol) or anti-diarrheal drug (loperamide) according to transit subtype for one month, antidepressants for 2 months, probiotics (ALFLOREX, SMEBIOCTA, PROBIOLOG FLORVIS) for 1 month, hypnosis for 5 hypnosis sessions in two months, Cognitive Behavioral Therapies for 2 months, colestyramine for IBS-D patients for 1 month, ondansetron for IBS-D patients and for 1 month, ebastine for 2 months, L-glutamine (5g x3/day, for 2 months, Gelsectan for one month, Biofeedback for 15 sessions in IBS-C (3 months), Low FODMAP diet for 1 month, gluten free diet for 1 month, standard dietary advice from the NICE (UK) for 1 month, increase in physical activity.
* Patient with health insurance (AME excepted)
* Informed written consent
* For women with childbearing potential, efficient contraception for the duration of the participation to the study

Exclusion Criteria:

* Other chronic gastrointestinal disease (celiac disease, inflammatory bowel disease)
* participants if there is a reason to suspect an alternative diagnosis to the IBS complaints
* Surgical intervention in the gastrointestinal region except for appendectomy, hernia repair, cholecystectomy and hemorroidectomy
* Treatment preceding FMT with: antibiotics, antifungic or probiotics treatment < 4 weeks, or factors that may affect the composition of intestinal microbiota
* Abuse of alcohol or drugs
* Pregnancy or breastfeeding
* Participation in any other interventional study
* Patients under legal protection.
* Acute COVID-19 infection
* Presence of systemic disease, immune deficiency or treatment with immune-modulators
* Severe psychiatric disorder
* Participants who were assessed as likely to be noncompliant (ie, not adhering to the tasks they were to perform as participants)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-07-15 (Estimated); Study Completion 2029-07-15 (Estimated)

PRIMARY OUTCOMES:
Decrease in IBS severity at 12 weeks defined by the percentage of patients having at least a 75 points decrease in IBS-SSS. | At 12 weeks
  To evaluate the efficacy of oral capsules containing frozen fecal microbiota (FMT) vs sham FMT on IBS severity score at 12 weeks in patients with irritable bowel syndrome with severe disease refractory to conventional treatments.
  Decrease in IBS severity at 12 weeks is defined by the percentage of patients having at least a 75 points decrease in IBS-SSS.

SECONDARY OUTCOMES:
Decrease in IBS severity at 12 weeks defined by the percentage of patients having at least a 50 points decrease in IBS-SSS. | At 12 weeks
  To evaluate the efficacy of oral capsules containing frozen fecal microbiota (FMT) vs sham FMT on IBS severity score at 12 weeks in patients with irritable bowel syndrome with severe disease refractory to conventional treatments (at least a 50 points decrease in IBS-SSS)
FMT success | At 12 weeks
  patient's microbiota 12 weeks after FMT closer to that of the donor than the patient's microbiota before FMT. The composition of the patient's fecal microbiota 12 weeks after FMT will be compared to the patient's microbiota before transplantation and to the donor using the Sorensen similarity index. The FMT will be considered as a success if the Sorensen index [patient after FMT vs donor] > Sorensen index [patient after FMT vs patient before FMT] and if the Sorensen index [patient after FMT vs donor] ≥ 0,6. The composition of fecal microbiota will be measured by pyrosequencing (16S RNA).
Intestinal microbiota composition at week 12 and 24 by 16s sequencing. | at week 12 and 24
  Intestinal microbiota composition and diversity at week 12 and 24 assessed by 16s sequencing. Microbiota composition and diversity assessed by 16s sequencing at week 12 and 24, compared to baseline and to healthy volunteers donor's microbiota. Microbiota composition will be assessed using Qiime pipeline and analyzed at all phylogenetic levels.
  Diversity will be evaluated using Shannon index, Simpson index, Chao1 index and number of observed species.
Efficacy (decrease in IBS severity >75 points) at week 24 according to FMT success. | At 24 weeks
  Efficacy (decrease in IBS severity >75 points) according to FMT success.
EMA Endpoint at week 12 and 24 defined as a patient who fulfils the response criteria (simultaneous improvement of transit and abdominal pain) displayed in the following for at least 50% of the observation time. | at week 12 and 24
  Efficacy according to EMA (European Medical Agency) endpoint in IBS on composite criteria at 12 or 24 weeks
Percentage of responders in the different subgroups IBS-D, IBS-C and IBS-M using the primary endpoint at week 12 and 24. | at week 12 and 24
  IBS severity at 12 weeks by donors (one donor giving FMT to several patients)
Mean IBS-SSS (IBS severity), comparison between FMT and placebo at 12 and 24 weeks) | at week 12 and 24
  IBS severity at 12 weeks and at 24 weeks by IBS subtypes according to transit pattern.
  The score ranges from 0 to 500 ( Remission : 0 to 74, Mild : 75 to 175, Moderate : 175 to 300 and Severe : >300).
Mean IBS-QoL score (IBS Quality of life) comparison between FMT and placebo at 12 and 24 weeks (Drossman et al. 2000) | at week 12 and 24
  IBS Quality of life at 12 weeks and 24 weeks. Irritable Bowel Syndrom- Quality of Life (IBS-QoL) at 12 weeks and 24 weeks, IBS-QoL ranges from 0 ( worse) to 100 (better).
Patient's perception of FMT : - Questionnaire for correct assessment of FMT or placebo and FMT acceptability) at V2 (FMT administration). - Questionnaire for assessment of FMT secondary effects at V3. | V2: five weeks after inclusion. V3:Four weeks after V2
  Patient's perception of FMT (questionnaire for correct assessment of FMT or placebo and FMT acceptability) (Annex D), secondary effects of FMT
Safety (Serious Adverse Events, Adverse Events) compared between groups. | through study completion, at 24 months
  Safety (Serious Adverse Events, Adverse Events) compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc SABATE, Pr, Study Director — Assistance Publique Hopitaux de Paris
Locations (1):
- Gastro-enterology department, Avicenne Hospital, Bobigny, France